CLINICAL TRIAL: NCT00540033
Title: Phase 2 Study of Oral Probiotics Reduce the Incidence and Severity of Necrotizing Enterocolitis for Very Low Birth Weight Infants -Multi-Center Randomized Control Trial
Brief Title: Probiotics Reduce Incidence of Necrotizing Enterocolitis for Very Low Birth Weight Infants
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: terminated because of enough case number
Sponsor: China Medical University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DMR94-IRB-14
Record Dates: First submitted 2007-10-03; First posted 2007-10-05 (Estimated); Last update posted 2007-10-05 (Estimated); Status verified 2007-10

CONDITIONS: Enterocolitis, Necrotizing
Keywords: probiotics; necrotizing enterocolitis; preterm very low birth weight infants (VLBW)
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2 (Experimental): Study arm was fed with probiotics as infloran 125mg/kg/dose twice daily by adding it to breast milk or mixed feeding (breast and formula) for 6 weeks; the control arm was fed with breast milk or mixed feeding without probiotics.
  Interventions: Dietary Supplement: infloran

INTERVENTIONS:
Dietary Supplement: infloran — Study group was fed with probiotics as infloran 125mg/kg/dose twice daily by adding it to breast milk or mixed feeding (breast and formula) for 6 weeks;
Dietary Supplement: infloran — Study group was fed with infloran [Lactobacilli acidophilus (CFU 109 NCDO 1748, obtained from the National Collection of Dairy Organisms)] and Bifidobacteria bifidum [(CFU 109, NCDO 1453 obtained from the National Collection of Dairy Organisms)]; Laboratorio Farmaceutico S.I.T S.r.I ITALY] 125mg/kg/dose twice daily by adding it to breast milk or mixed feeding (breast and formula) for 6 weeks;

SUMMARY:
We investigate the efficacy of probiotics in reducing the incidence and severity of necrotizing enterocolitis (NEC) for very low birth weight (VLBW) infants.A prospective, masked, multi-center randomized control trial will be conducted level III neonatal center to evaluate the beneficial effects of probiotics for NEC among VLBW (<1500 g) infants. VLBW infants who start to feed enterally are eligible and are randomized into 2 groups after parental informed consents were obtained. Infants in the study group are fed with Infloran (Lactobacillus acidophilus and Bifidobacterium bifidus) with breast or formula milk twice daily for 6 weeks. Infants in the control group are fed with breast or formula milk alone. The clinicians caring for the infants are blinded to the group assignment. The primary outcome measurement is death or NEC (≧stage 2).

DETAILED DESCRIPTION:
Introduction NEC is a worldwide problem in preterm very low birth weight (VLBW) infants with highly variable incidence affecting 2.6% to 28% of these infants; 1.2.Recent reports suggest increasing occurrence of NEC, estimating up to 9000 cases of NEC in the United States every year, with death occurring in 20 % to 40% of affected individuals. [1.3] As the number of very low-birth-weight infants increases, NEC remains a critical eminent problem. 3[4] The pathogenesis of NEC is unknown, but is widely considered as a multi-factorial disease; prematurity, enteral feeding, intestinal hypoxia-ischemia, and bacterial colonization are considered major risk factors. [4] Researches showed that proinflammatory cytokines, such as interleukin-1.6.8. (IL-1, IL-6, IL-8) and tumor necrosis factor- (TNF- ) 5-711-13 and anti-inflammatory cytokines such as IL-10 and transforming growth factor- (TGF- ) 8-1014-16 by intestinal epithelial cells is highly relevant to be involved in the final common pathway of pathogen of NEC.5-10 11-16.In mature bowel, the intestinal environment is capable of producing an array of cytokines important in the development and control of inflammatory responses11 8. In contrast, the immaturity of the neonatal intestinal immune system is evidenced by decreased numbers of immune cells 12.13 9.10. Recently, it has bee thought that inappropriate, accentuated inflammatory response to colonizing pathogenic flora at premature gut plays a major role, the inflammatory cascade further promotes spread of bacteria or toxin, and end up with ischemia, necrosis and even perforation. 14-1617.18.19 We and Bin-Nun had proved that probitics reduces the incidence and severity of necrotizing enterocolitis in preterm VLBW infants. 17.18 Nevertheless, there is no solid data in the literature as to the optima strains, timing, dosage and duration of probiotics administering to preterm VLBW infants at preset; and these need further investigate.

Bifidobacteria and lactobacilli are commonly found in breast-fed infants; 19 and most of the NEC in VLBW infants occurred before 6-8 weeks of age; 20 therefore, we hypothesized that early oral probiotics contains Bifidobacteria and lactobacilli fed to preterm VLBW infants for 6 weeks could reduce the incidence and severity of NEC.

PATIENTS AND METHODS From July 1, 2005 to Dec 31, 2006, a prospective masked randomized control trial will be conducted at the level III Neonatal Intensive Care Unit (NICU) of eight neonatal centers in Taiwan. Study is approved by Institutional Review Board (IRB) of each hospital. Preterm VLBW infants (birth weight < 1500 gm) who were enterally fed are eligible for the trial. They are randomized into the study or control group by a random number table sequence after informed parental consents were obtained. The allocations are contained in opaque sequentially numbered and sealed envelopes. Preterm VLBW infants who have severe asphyxia (stage III), fetal chromosome anomalies, fetal cyanotic congenital heart disease, congenital intestine atresia, gastroschisis and omphalocele were excluded.

The clinicians who provided care to the infants are blinded to the grouping. Investigators were not involved in the care of these infants. Study group is fed with infloran (Lactobacillus acidophilus and Bifidobacterium bifidus, Swiss Serum and Vaccine Institute Berne, Switzerland) 125mg/kg/dose (CFU 109) twice daily with breast milk for 6 weeks; the control group is fed with breast milk alone. Infloran was stored in refrigerator at a tempreture between 2 -80 C and mixed with breast milk before feeding. Breast milk was either from infant's own mother's milk or from breast milk bank. Both breast milk of the study and control group are prepared by breast milk team who were not involved in the care of the infant and follow the order from a sealed envelop. Feeding is started when the infant*s vital signs were stable, have active bowel movement, without abdominal distension, without bile or blood from the nasogastric tube, and did not have an umbilical artery or umbilical venous catheter in place for at least 24 hours.

A strict feeding protocol is followed for all study infants. Depending on the birth weight and gestational age, a certain amount of breast milk is initiated after the infant tolerated one trial of distilled water. On the first day, 1 mL/kg - distilled water was given twice, followed by breast milk. The amount of feeding was advanced slowly if tolerated, with no more than 20 mL/kg/day of increment per feed. An oral intake of 100 mL/kg/d is defined as complete enteral feeding. Feeding was stopped if there was any sign of feeding intolerance, defined as the presence of gastric aspirate in the amount that was more than half of the previous feeding, twice, with abdominal distension. Infants who weighed under 1,000gm received total parenteral nutrition (TPN) until half of the calories were supplied by oral route. The same attending physician is in charge of the care of the infants during their hospital stay. The residents who rotated through the NICU provided the care following established protocols in the unit. Definition of prenatal steroid, small for gestational age, prolonged rupture of amniotic membrane, chorioamnionitis, asphyxia, respiratory distress syndrome, patent ductus arteriosus, intraventricular hemorrhage (IVH), sepsis; indication of surfactant and indomethacin are described as in our previous study. [16 ] There were no modifications in any management protocols, clinical practices, equipment, infrastructure, or any other elements in the unit during the study period, and all the protocols got consensus in the eight centers after several discussion.

NEC is classified by modified Bell's classification. 21[39] The final determination of the diagnosis of NEC (≧ stage2) is made by two independent attending physicians who did not know the group assignment of the infant. Demographic and clinical variables that are potential risk factors for NEC were prospectively abstracted from the medical records. These factors included chorioamnionitis, prolonged rupture of amniotic membrane (PROM) >18 hours, pre-eclampsia, use of prenatal steroid, multiple -pregnancy, mode of delivery, gender, gestational age, birth weight, small for gestational age, Apgar score at 5 minutes, asphyxia, initial Hb, initial body temperature, use of surfactant, use of indomethacin, dosage of indomethacin, days of UAC and UVC, days of fasting, use of dopamine, days of antibiotics use, days of dopamine use, incidence and grading of IVH, incidence of pneumothorax, days of mechanical ventilation and oxygen supplement, days of TPN before and after NEC; weight gain per week, lengthy of stay are prospectively abstracted from the medical records.

Primary outcome measurement was the incidence and severity of NEC (≧ stage2); and death. Secondary outcome were, culture proved sepsis, chronic lung disease, periventricular leukomalacia (PVL) , weight gain per week, duration of TPN, lengthy of stay, cost effective analysis.

SAMPLE SIZE CALCULATION AND STATISTICS According to the unpublished data of Premature Baby Foundation of Taiwan and Bravura of National Health Insurance (2003-2004), the recent data showed that the combined incidence of NEC (≧stage 2) or death for preterm VLBW infants was about 25 % for level III neonatal center in Taiwan. Setting the α error at 0.05 and β error at 0.1; and an absolute reduction of the incidence of NEC or death by 50%, the number needed to verify our hypothesis was 203 for each arm.

ELIGIBILITY:
Inclusion Criteria:

* Preterm VLBW infants (birth weight < 1500 gm) who are enterally fed are eligible for the trial.

Exclusion Criteria:

* Preterm VLBW infants who have severe asphyxia (stage III), fetal chromosome anomalies, fetal cyanotic congenital heart disease, congenital intestine atresia, gastroschisis and omphalocele are excluded.

Ages: 1 Day to 3 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 217 (Actual)
Dates: Start 2005-02; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome measurement was death or NEC (≧stage 2) | From April 1, 2005 to May 30, 2007

SECONDARY OUTCOMES:
Secondary outcome were culture proved sepsis, chronic lung disease, periventricular leukomalacia (PVL) , weight gain per week, duration of TPN, lengthy of stay, cost effective analysis. | From April 1, 2005 to May 30, 2007,

CONTACTS AND LOCATIONS:
Overall Officials: HUNG-CHIH LIN, MD, Study Chair — Department of Pediatrics, Children Hospital, China Medical University, Taichung, Taiwan
Locations (1):
- Department of Pediatrics, Children Hospital, China Medical University, Taichung, Taiwan, Taichung, Taichung,, Taiwan

REFERENCES:
- [Derived] Lin HC, Hsu CH, Chen HL, Chung MY, Hsu JF, Lien RI, Tsao LY, Chen CH, Su BH. Oral probiotics prevent necrotizing enterocolitis in very low birth weight preterm infants: a multicenter, randomized, controlled trial. Pediatrics. 2008 Oct;122(4):693-700. doi: 10.1542/peds.2007-3007. PMID 18829790